CLINICAL TRIAL: NCT04654260
Title: Behavior Therapy for Irritability and Aggression in Adolescents With Autism
Brief Title: Behavior Therapy for Irritability in Autism
Acronym: BTIA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0102012121-5; W81XWH2010718 (Other Grant/Funding Number: DoD, Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2020-12-02; First posted 2020-12-04 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder; Irritability; Disruptive Behavior; Anger; Aggression; Asperger Syndrome; Pervasive Developmental Disorder
Keywords: autism; adolescents; behavior therapy; treatment; disruptive behavior; irritability; anger; aggression
MeSH Terms: conditions — Autism Spectrum Disorder; Problem Behavior; Aggression; Asperger Syndrome; Child Development Disorders, Pervasive; Autistic Disorder | interventions — Behavior Therapy; Palliative Care

STUDY DESIGN:
Intervention Model Description: This is randomized controlled trial of behavior therapy for irritability versus a supportive therapy control condition
Who Masked: Outcomes Assessor
Masking Description: Primary outcomes will be assessed by an independent evaluator who will be "blinded" to subject's treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Therapy for Irritability in Autism (BTIA) (Experimental): BTIA consists of 15 ninety-minute weekly sessions that will be conducted with the teens and their parents by experienced therapists using a structured, detailed manual.
  Interventions: Behavioral: Behavioral Therapy for Irritability in Autism
- Psychoeducation and Supportive Therapy (PST) (Active Comparator): PST consist of 15 weekly, ninety-minute sessions focused on learning about and discussing issues of diagnosis, treatment and educational services with an experienced therapist could be helpful to children on the autism spectrum and their families.
  Interventions: Behavioral: Psychoeducation and Supportive Therapy (PST)

INTERVENTIONS:
Behavioral: Behavioral Therapy for Irritability in Autism — The child-focused components of BTIA are organized in modules dedicated to emotion regulation, problem solving and practice of planned steps to prevent or resolve conflicts. Each session contains a set of six to seven goals, and each goal contains a menu of techniques and activities that can be used to attain this goal. In order to administer the treatment in a flexible yet reliable manner, the therapist works collaboratively with the child and his or her parents to select activities that are perceived as relevant for attaining the session's goal. The parent-focused components of BTIA include include education about the effects of antecedents and consequences on disruptive behavior, developing strategies for reducing or altering antecedent events that may lead to disruptive reactions and helping parents to use reinforcement of competent and calm responses in potentially frustrating situations.
  Arms: Behavioral Therapy for Irritability in Autism (BTIA)
Behavioral: Psychoeducation and Supportive Therapy (PST) — Each PST session will start with a review of events of the past week and include queries of topics such as school, interests, hobbies, and family with an overarching goal of enhancing subjective well-being. A major objective is to enables the participant to discuss his or her concerns with a therapist toward a goal of enhancing overall psychological wellbeing. Education about autism diagnosis and services is also provided to families as part of PST.
  Arms: Psychoeducation and Supportive Therapy (PST)

SUMMARY:
This is a clinical trial of a novel intervention, Behavioral Therapy for Irritability and Aggression (BTIA), for adolescents on the autism spectrum. The main goals of BTIA are to help adolescents develop emotion regulation skills to handle frustration and to strengthen skills for navigating the challenging and diverse experiences associated with the transition to adulthood. The study will test whether BTIA can be helpful to adolescents on the autism spectrum and to their families.

DETAILED DESCRIPTION:
This is a randomized controlled study of BTIA versus a supportive therapy control condition in 126 adolescents (ages 12 to 18 years) with a diagnosis of autism spectrum disorder and significant levels of disruptive behaviors such as aggression, anger outbursts, and oppositional behavior. BTIA consists of 15 ninety-minute weekly sessions that will be conducted with the teens and their parents by therapists using a structured, detailed manual. The effects of BTIA on the reduction of behavioral problems will be rated by an experienced clinician who does not know which treatment each participant is receiving (a "blinded" evaluator). Study participants will receive a thorough diagnostic assessment of autism spectrum disorder and other forms of psychopathology that may co-occur with ASD. In addition to testing the effects of BTIA on disruptive behavior, the changes in adaptive functioning, or children's ability to function competently in their everyday environment, will be examined before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls, ages 12 to 18 years inclusive
* Diagnosis of autism spectrum disorder
* Presence of disruptive behaviors such as irritability and anger outbursts
* No planned changes in the intensity of current treatment(s)
* Medication free or on stable medication
* Sufficient language for participation in verbal therapy
* Lives within driving distance from New Haven, CT

Exclusion Criteria:

* Presence of a medical condition that would interfere with participation in the study
* Presence of a current psychiatric disorder that requires immediate clinical attention

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Modified Overt Aggression Scale (MOAS) | baseline (week 0)
  Modified Overt Aggression Scale is a 16-item scale that reflects the frequency and severity of incidents of aggressive behavior. Scores can range from 0 (minimum) to 300 (maximum) with higher scores reflecting worse outcome.
Modified Overt Aggression Scale (MOAS) | midpoint (week 8)
  Modified Overt Aggression Scale is a 16-item scale that reflects the frequency and severity of incidents of aggressive behavior. Scores can range from 0 (minimum) to 300 (maximum) with higher scores reflecting worse outcome.
Modified Overt Aggression Scale (MOAS) | endpoint (week 16)
  Modified Overt Aggression Scale is a 16-item scale that reflects the frequency and severity of incidents of aggressive behavior. Scores can range from 0 (minimum) to 300 (maximum) with higher scores reflecting worse outcome.
Modified Overt Aggression Scale (MOAS) | six-month follow up (week 42)
  Modified Overt Aggression Scale is a 16-item scale that reflects the frequency and severity of incidents of aggressive behavior. Scores can range from 0 (minimum) to 300 (maximum) with higher scores reflecting worse outcome.
The Clinical Global Impression - Improvement Score (CGI-I) | baseline (week 0)
  The Clinical Global Impression - Improvement Score assigned by an independent evaluator (IE) who will be blind to treatment assignment is the categorical primary outcome measure of aggressive behavior. The CGI-I reflects the IE's assessment of overall change from baseline rated on a scale from 1 to 7 where 1 is very much improved, 2 is much improved, 3 is minimally improved, 4 is no change, 5 is minimally worse, 6 is much worth, and 7 is very much worse. Higher scores reflect worse outcome. By convention, ratings of very much improved (1) or much improved (2) define positive response; all other scores are classified as a negative response.
The Clinical Global Impression - Improvement Score (CGI-I) | midpoint (week 8)
  The Clinical Global Impression - Improvement Score assigned by an independent evaluator (IE) who will be blind to treatment assignment is the categorical primary outcome measure of aggressive behavior. The CGI-I reflects the IE's assessment of overall change from baseline rated on a scale from 1 to 7 where 1 is very much improved, 2 is much improved, 3 is minimally improved, 4 is no change, 5 is minimally worse, 6 is much worth, and 7 is very much worse. Higher scores reflect worse outcome. By convention, ratings of very much improved (1) or much improved (2) define positive response; all other scores are classified as a negative response.
The Clinical Global Impression - Improvement Score (CGI-I) | endpoint (week 16)
  The Clinical Global Impression - Improvement Score assigned by an independent evaluator (IE) who will be blind to treatment assignment is the categorical primary outcome measure of aggressive behavior. The CGI-I reflects the IE's assessment of overall change from baseline rated on a scale from 1 to 7 where 1 is very much improved, 2 is much improved, 3 is minimally improved, 4 is no change, 5 is minimally worse, 6 is much worth, and 7 is very much worse. Higher scores reflect worse outcome. By convention, ratings of very much improved (1) or much improved (2) define positive response; all other scores are classified as a negative response.
The Clinical Global Impression - Improvement Score (CGI-I) | six-month follow up (week 42)
  The Clinical Global Impression - Improvement Score assigned by an independent evaluator (IE) who will be blind to treatment assignment is the categorical primary outcome measure of aggressive behavior. The CGI-I reflects the IE's assessment of overall change from baseline rated on a scale from 1 to 7 where 1 is very much improved, 2 is much improved, 3 is minimally improved, 4 is no change, 5 is minimally worse, 6 is much worth, and 7 is very much worse. Higher scores reflect worse outcome. By convention, ratings of very much improved (1) or much improved (2) define positive response; all other scores are classified as a negative response.
Irritability subscale - Aberrant Behavioral Checklist | baseline (week 0)
  The 15-item Irritability subscale includes questions about aggression, tantrums, agitation, and unstable mood that are rated on a 4-point scale with the following anchor points: 0 = not at all a problem; 1 = the behavior is a problem but slight in degree; 2 = the problem is moderately serious; 3 = the problem is severe in degree. The total Irritability subscale score ranges from 0 to 45, with higher scores indicating greater severity.
Irritability subscale - Aberrant Behavioral Checklist | midpoint (week 8)
  The 15-item Irritability subscale includes questions about aggression, tantrums, agitation, and unstable mood that are rated on a 4-point scale with the following anchor points: 0 = not at all a problem; 1 = the behavior is a problem but slight in degree; 2 = the problem is moderately serious; 3 = the problem is severe in degree. The total Irritability subscale score ranges from 0 to 45, with higher scores indicating greater severity.
Irritability subscale - Aberrant Behavioral Checklist | endpoint (week 16)
  The 15-item Irritability subscale includes questions about aggression, tantrums, agitation, and unstable mood that are rated on a 4-point scale with the following anchor points: 0 = not at all a problem; 1 = the behavior is a problem but slight in degree; 2 = the problem is moderately serious; 3 = the problem is severe in degree. The total Irritability subscale score ranges from 0 to 45, with higher scores indicating greater severity.
Irritability subscale - Aberrant Behavioral Checklist | six-month follow up (week 42)
  The 15-item Irritability subscale includes questions about aggression, tantrums, agitation, and unstable mood that are rated on a 4-point scale with the following anchor points: 0 = not at all a problem; 1 = the behavior is a problem but slight in degree; 2 = the problem is moderately serious; 3 = the problem is severe in degree. The total Irritability subscale score ranges from 0 to 45, with higher scores indicating greater severity.

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scales - Communication Domain Score | baseline (week 0)
  Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) is a measure of competence in communication, daily living skills, and socialization which is administered in a semi-structured parent interview format. Items assess the individual's behavior in these domains and are rated according to the frequency with which behaviors are performed without help or prompting (i.e., "Never," "Sometimes" or "Usually"). The raw scores are converted to standard scores (mean = 100, SD = 15; range 40 to 160), and higher scores indicate better adaptive functioning.
Vineland Adaptive Behavior Scales - Communication Domain Score | endpoint (week 16)
  Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) is a measure of competence in communication, daily living skills, and socialization which is administered in a semi-structured parent interview format. Items assess the individual's behavior in these domains and are rated according to the frequency with which behaviors are performed without help or prompting (i.e., "Never," "Sometimes" or "Usually"). The raw scores are converted to standard scores (mean = 100, SD = 15; range 40 to 160), and higher scores indicate better adaptive functioning.
Vineland Adaptive Behavior Scales - Communication Domain Score | six-month follow up (week 42)
  Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) is a measure of competence in communication, daily living skills, and socialization which is administered in a semi-structured parent interview format. Items assess the individual's behavior in these domains and are rated according to the frequency with which behaviors are performed without help or prompting (i.e., "Never," "Sometimes" or "Usually"). The raw scores are converted to standard scores (mean = 100, SD = 15; range 40 to 160), and higher scores indicate better adaptive functioning.

OTHER OUTCOMES:
Affective Reactivity Index (ARI) | baseline (week 0)
  Affective Reactivity Index (ARI) is an 7-item measure of anger and irritability in children and adolescents which is reliable in ASD. Items are scored of a 0, 1 or 3 scale and first 6 items are summed for a total score, with a possible range from 0 to 12, higher scores reflecting greater levels of irritability
Affective Reactivity Index (ARI) | midpoint (week 8)
  Affective Reactivity Index (ARI) is an 7-item measure of anger and irritability in children and adolescents which is reliable in ASD. Items are scored of a 0, 1 or 3 scale and first 6 items are summed for a total score, with a possible range from 0 to 12, higher scores reflecting greater levels of irritability
Affective Reactivity Index (ARI) | endpoint (week 16)
  Affective Reactivity Index (ARI) is an 7-item measure of anger and irritability in children and adolescents which is reliable in ASD. Items are scored of a 0, 1 or 3 scale and first 6 items are summed for a total score, with a possible range from 0 to 12, higher scores reflecting greater levels of irritability
Affective Reactivity Index (ARI) | six-month follow up (week 42)
  Affective Reactivity Index (ARI) is an 7-item measure of anger and irritability in children and adolescents which is reliable in ASD. Items are scored of a 0, 1 or 3 scale and first 6 items are summed for a total score, with a possible range from 0 to 12, higher scores reflecting greater levels of irritability
Social Responsiveness Scale-2 (SRS-2) | baseline (week 0)
  Social Responsiveness Scale-2 (SRS-2) is a 65-item, parent-report scale that measures social disability. Items assess the individual's social awareness, social cognition, social communication, social motivation, and restricted interest and repetitive behaviors on a scale from 0 to 3. The raw scores are converted to T-scores (mean = 50, SD = 10; range 30 to 90), and higher scores indicate greater impairment.
Social Responsiveness Scale-2 (SRS-2) | midpoint (week 8)
  Social Responsiveness Scale-2 (SRS-2) is a 65-item, parent-report scale that measures social disability. Items assess the individual's social awareness, social cognition, social communication, social motivation, and restricted interest and repetitive behaviors on a scale from 0 to 3. The raw scores are converted to T-scores (mean = 50, SD = 10; range 30 to 90), and higher scores indicate greater impairment.
Social Responsiveness Scale-2 (SRS-2) | endpoint (week 16)
  Social Responsiveness Scale-2 (SRS-2) is a 65-item, parent-report scale that measures social disability. Items assess the individual's social awareness, social cognition, social communication, social motivation, and restricted interest and repetitive behaviors on a scale from 0 to 3. The raw scores are converted to T-scores (mean = 50, SD = 10; range 30 to 90), and higher scores indicate greater impairment.
Social Responsiveness Scale-2 (SRS-2) | six-month follow up (week 42)
  Social Responsiveness Scale-2 (SRS-2) is a 65-item, parent-report scale that measures social disability. Items assess the individual's social awareness, social cognition, social communication, social motivation, and restricted interest and repetitive behaviors on a scale from 0 to 3. The raw scores are converted to T-scores (mean = 50, SD = 10; range 30 to 90), and higher scores indicate greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Sukhodolsky, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Research data from this study will be shared via the National Database for Autism Research and NIH Data Repositories (https://nda.nih.gov/) consistent with the Yale University Policy. The data management for this study will be conducted using the OnCore system at YCCI (https://medicine.yale.edu/ycci/oncore/), which enables translation of data to de-identified data sets that can be placed online using GUID technology as specified in Federal guidelines. At the time of permission/consent/assent, participants and their parents will be informed of the data-sharing plan. Raw data generated by the project will be quality-certified by our research team (including fidelity to research procedures, proper file format, artifact removal, and de-identifying, resulting in artifact-free raw data) prior to submission to NDAR for usability. Consistent with the NDAR data sharing policy, data will be submitted, at the individual level, on all enrolled subjects.
Supporting Information: Study Protocol, SAP
Time Frame: Analyzed data will be submitted at the time of publication, and publications resulting from these data will be associated with NDAR entries using the NDAR Study Feature.
Access Criteria: Data generated with funds from this grant will be freely available on the NIH/NDAR database

REFERENCES:
- [Background] Sukhodolsky DG, Smith SD, McCauley SA, Ibrahim K, Piasecka JB. Behavioral Interventions for Anger, Irritability, and Aggression in Children and Adolescents. J Child Adolesc Psychopharmacol. 2016 Feb;26(1):58-64. doi: 10.1089/cap.2015.0120. Epub 2016 Jan 8. PMID 26745682
- [Background] Scahill L, Bearss K, Lecavalier L, Smith T, Swiezy N, Aman MG, Sukhodolsky DG, McCracken C, Minshawi N, Turner K, Levato L, Saulnier C, Dziura J, Johnson C. Effect of Parent Training on Adaptive Behavior in Children With Autism Spectrum Disorder and Disruptive Behavior: Results of a Randomized Trial. J Am Acad Child Adolesc Psychiatry. 2016 Jul;55(7):602-609.e3. doi: 10.1016/j.jaac.2016.05.001. Epub 2016 May 7. PMID 27343887
- [Background] Ibrahim K, Eilbott JA, Ventola P, He G, Pelphrey KA, McCarthy G, Sukhodolsky DG. Reduced Amygdala-Prefrontal Functional Connectivity in Children With Autism Spectrum Disorder and Co-occurring Disruptive Behavior. Biol Psychiatry Cogn Neurosci Neuroimaging. 2019 Dec;4(12):1031-1041. doi: 10.1016/j.bpsc.2019.01.009. Epub 2019 Feb 4. PMID 30979647
- [Background] Ibrahim K, Kalvin C, Marsh CL, Anzano A, Gorynova L, Cimino K, Sukhodolsky DG. Anger Rumination is Associated with Restricted and Repetitive Behaviors in Children with Autism Spectrum Disorder. J Autism Dev Disord. 2019 Sep;49(9):3656-3668. doi: 10.1007/s10803-019-04085-y. PMID 31144231
- [Background] Henriksen M, Skrove M, Hoftun GB, Sund ER, Lydersen S, Tseng WL, Sukhodolsky DG. Developmental Course and Risk Factors of Physical Aggression in Late Adolescence. Child Psychiatry Hum Dev. 2021 Aug;52(4):628-639. doi: 10.1007/s10578-020-01049-7. PMID 32852728
- [Background] Kalvin CB, Gladstone TR, Jordan R, Rowley S, Marsh CL, Ibrahim K, Sukhodolsky DG. Assessing Irritability in Children with Autism Spectrum Disorder Using the Affective Reactivity Index. J Autism Dev Disord. 2021 May;51(5):1496-1507. doi: 10.1007/s10803-020-04627-9. PMID 32734421